CLINICAL TRIAL: NCT03501264
Title: Evaluation of an Online Intervention to Help LGBTQ Youth Cope With Bullying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Egan, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO17060347; 5R21HD083561-02 (NIH)
Record Dates: First submitted 2018-03-13; First posted 2018-04-18 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Bullying of Child

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group receives the game
  Interventions: Behavioral: Online Game
- Control Group (Active Comparator): This group receives LGBTQ resources only
  Interventions: Behavioral: LGBTQ Resources

INTERVENTIONS:
Behavioral: Online Game — LGBTQ Bullying game
  Arms: Intervention group
Behavioral: LGBTQ Resources — This group receives LGBTQ Resources
  Arms: Control Group

SUMMARY:
The purpose of this research study is to conduct a pilot randomized controlled trial of a game-based intervention is able to increase help-seeking-related knowledge, attitudes, and behaviors, reduce health risk factors/behaviors, and increase resiliencies among sexual and gender minority (SGM) youth. The goals of the proposed study are to: (1) Test the feasibility and acceptability of a game-based intervention to increase help-seeking-related knowledge, attitudes, and behaviors among SGM youth; and (2) Using a randomized controlled trial, test the efficacy of a game-based intervention to increase help-seeking-related knowledge, attitudes, and behaviors, reduce health risk factors/behaviors, and increase resiliencies among SGM youth.

DETAILED DESCRIPTION:
The purpose of this research study is to conduct a pilot randomized controlled trial of a game-based intervention is able to increase help-seeking-related knowledge, attitudes, and behaviors, reduce health risk factors/behaviors, and increase resiliencies among sexual and gender minority (SGM) youth. The goals of the proposed study are to: (1) Test the feasibility and acceptability of a game-based intervention to increase help-seeking-related knowledge, attitudes, and behaviors among SGM youth; and (2) Using a randomized controlled trial, test the efficacy of a game-based intervention to increase help-seeking-related knowledge, attitudes, and behaviors, reduce health risk factors/behaviors, and increase resiliencies among SGM youth.

ELIGIBILITY:
Inclusion Criteria:

* Must identify as lesbian, gay, bisexual, queer, transgender or another sexual or gender minority
* must have bullying experience
* must have access to a computer and email

Exclusion Criteria:

* Residence outside of United States
* Not within the age range

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Egan, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Coulter RW, Sang JM, Louth-Marquez W, Henderson ER, Espelage D, Hunter SC, DeLucas M, Abebe KZ, Miller E, Morrill BA, Hieftje K, Friedman MS, Egan JE. Pilot Testing the Feasibility of a Game Intervention Aimed at Improving Help Seeking and Coping Among Sexual and Gender Minority Youth: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Feb 15;8(2):e12164. doi: 10.2196/12164. PMID 30767903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 120 | 120
Completed | 120 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Customized [Count of Participants; unit: Participants] — Years Old
  Participants
    14 | 16 | 19 | 35
    15 | 33 | 33 | 66
    16 | 37 | 34 | 71
    17 | 28 | 28 | 56
    18 | 6 | 6 | 12
Sex/Gender, Customized [Count of Participants; unit: Participants]
  cisgender boys | 18 | 21 | 39
  cisgender girls | 39 | 49 | 88
  gender minority | 63 | 50 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 21 | 49
  Not Hispanic or Latino | 92 | 99 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 5 | 8
  Black or African American | 9 | 3 | 12
  White | 86 | 85 | 171
  More than one race | 14 | 19 | 33
  Unknown or Not Reported | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Help Seeking Scores
Description: A measure of help-seeking intentions for emotional/mental distress from different sources of help. Options range from 1= never, 2=rarely, 3=occasionally, 4=a moderate amount, 5=a great deal. Total scale is out of 105 with higher scores indicating greater health seeking intentions. Questions were asked about: parents/guardians, relatives/family member, teacher, friend, mental health professional, nurse or doctor, and phone/chat line. Mean scores will be calculated at baseline and 1-month post intervention. These scores will then be compared to determine change over the intervention period.
Time Frame: Baseline and 1-month post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 72 | 83
Participants
  Positive Change - yes | 28 | 28
  Positive Change - no | 44 | 55

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT03501264/Prot_SAP_000.pdf